CLINICAL TRIAL: NCT03948308
Title: Alteration of the Immune Response in Bacterial Infection
Acronym: ARIIBACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Roderick Meckenstock, Principal Investigator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P17/03_ARIIBACT
Record Dates: First submitted 2019-04-15; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): blood sample before, during and after treatment for infection
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — blood sample before, during and after infection treatment

SUMMARY:
The pilot study "ARIIBO" was conducted to analyze changes in immune parameters reported in obese subjects, which had never been the subject of a global study outside of an infectious context, and studied in period septic only sporadically. This study was intended to contribute to a better understanding of the probably adverse impact of obesity on the immune response to bacterial infections, and to describe a specific immunological profile of an infectious excess risk in obese subjects.

In terms of infection, obesity is a risk factor due to "mechanical" and pharmacodynamic variations, but also to the immune system. One of the best studied immunological parameters in obese patients, leptin resistance, is associated with a decrease in innate and adaptive immunity through a modification of the lymphocyte and cytokine profile.

It is important to compare the data collected in obese patients infected (first study called "ARIIBO"), with those of non-obese subjects presenting the same type of infection, which will be included in the study "ARIIBACT"

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* BMI 18 to 25
* presence of a bacterial infection
* pneumopathy (documented or probable)
* acute pyelonephritis / prostatitis
* skin and soft tissue infection (erysipelas, fasciitis, excluding pressure ulcers)
* cholecystitis / cholangitis,
* surgical site infection
* signed informed consent

Exclusion Criteria:

* patients with documented viral, parasitic or mycotic infections
* patients with bacterial infection> 4 weeks (eg endocarditis, osteoarticular infections)
* patients followed in intensive unit care
* patients with progressive cancerous pathology or malignant hemopathy diagnosed in the previous five years
* patients with systemic diseases (connective tissue diseases, vasculitis)
* known immunodepression syndrome (CVID, HIV ...)
* immunosuppressive therapy in progress until less than one month before inclusion (corticosteroids, DMARDs, biotherapies, hydroxychloroquine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
cytokin analysis (IL-6, IL-10, IL-17, TNFα, IFNγ) | 1 month
  Description of an immunological profile of inflammation using current inflammatory cytokines during sepsis in non-obese subjects in comparison with this same profile in obese subjects
adipokin analysis (leptine, adiponectine) | 1 month
  Description of the kinetics of 2 cytokines more speficically involved in obesity (leptine, adipokinine) during sepsis in non-obese subjects in comparison with this same profile in obese subjects
leptin polymorphism analysis | 1 month
  Description of the genetic polymorphism of leptine and leptine receptor in non-obese subjects in comparison with this same profile in obese subjects

CONTACTS AND LOCATIONS:
Locations (1):
- CH Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No